CLINICAL TRIAL: NCT05831319
Title: A Prospective, Multicenter, Observational Study Evaluating Standard of Care Practices, Procedural Outcomes, and In-hospital Complications of Endovascular Procedures for Treatment of Atherosclerotic Lesions in the Infrainguinal Arteries
Brief Title: Evaluation of Standard of Care Practices, Procedural Outcomes and In-hospital Complications of Peripheral Endovascular Procedures
Acronym: BIO-OSCAR SOC
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C2201
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Above the knee (ATK) group: Target lesions located in the superficial femoral artery or popliteal arteries (above the tibial plateau)
- Below the knee (BTK) group: Target lesions involve arteries below the tibial plateau

SUMMARY:
Significant advances in dedicated materials and techniques along with increased operator experience led to a significant increment in procedural success rate of peripheral endovascular interventions, exceeding 90% in expert hands with reported low procedural complication rates. However, there are still lack of data on procedural outcomes, in-hospital complications, and resource utilization on treatment of (complex) lesions in the femoral, popliteal and infrapopliteal artery in the real-world condition in Europe.

DETAILED DESCRIPTION:
The study will enroll consecutive eligible subjects who have peripheral artery disease (PAD) requiring endovascular treatment of de-novo and restenotic atherosclerotic lesions in femoral, popliteal and infrapopliteal arteries.

The purpose of this prospective, multicenter, observational European Study is to evaluate the standard of care practices, procedural outcomes, and in-hospital complications of endovascular peripheral interventions for treatment of lesions in the femoral, popliteal and infrapopliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥18 years old
2. Subject has provided written informed consent
3. Subject has Rutherford classification 2 to 6
4. Reference vessel diameter ≥2 and ≤7 mm
5. Target lesion(s) has stenosis >70% by visual assessment
6. Multiple consecutive single lesions with a healthy segment(s) of ≤ 3cm in-between the lesions will be considered one lesion.

   For Above the knee (ATK) group
7. Target lesions located in the superficial femoral artery or popliteal arteries (above the tibial plateau)
8. At least 1 below-knee artery patent to the ankle
9. Successful treatment of inflow iliac stenosis to the target lesion. Inflow lesion stenosis can be treated during the same procedure as per local standard of care.

   For Below the knee (BTK) group:
10. Target lesions involve arteries below the tibial plateau
11. Successful treatment of inflow vessel (from ipsilateral iliac to the target lesion) resulting in ≤30% residual stenosis with no evidence of embolization or significant complications.

Exclusion Criteria:

1. Subject has a single target lesion that involves both ATK and BTK segment.
2. Subject not suitable for receiving endovascular procedures of lower limb arteries
3. Prior planned major amputation in the target limb (above the ankle)
4. Subject with previous bypass surgery of target vessel.
5. History of any open surgical procedure within the past 30 days.
6. Planned vascular surgery procedure within the next 30 days after the ATK and/or BTK procedure on the target limb. Note: The inflow vessels can be treated on the day of the procedure
7. Subject under dialysis
8. Subject currently enrolled in another investigational device, biologic, or drug trial in which the primary endpoint has not yet been reached
9. Subject lacking capacity to provide informed consent
10. Subject under judicial protection, tutorship, or curatorship (for France only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have PAD with target lesion(s) located in the femoral, popliteal and/or infrapopliteal artery are eligible for the study. Up to 380 subjects will be enrolled in approximately 12 investigational sites in Europe.
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Procedural success rate | Index Procedure
  Combination of technical success and absence of procedural complications

SECONDARY OUTCOMES:
Procedure technical success rate | Index Procedure
  successful crossing and achievement of a final residual diameter stenosis of ≤30% of the treated target lesion on the procedural completion angiography
Rate of target lesion bailout stenting | Index Procedure
  Stented target lesion
Stented length | Index Procedure
  Stented length
Rate of PTA balloon related flow-limiting dissections | Index Procedure
  PTA balloon related flow-limiting dissections
Rate of distal embolization | Index Procedure
  Distal embolization
Rate of target vessel rupture | Index Procedure
  Target vessel rupture
Rate of target vessel perforation | Index Procedure
  Target vessel perforation
Rate of acute occlusion | Index Procedure
  Acute occlusion
Primary crossing success rate | Index Procedure
  Successfully placement of a guidewire into the distal true lumen with the primary crossing strategy
Rate of Serious Adverse Device Effects | Index Procedure
  Serious Adverse Device Effects
Non-labor resource use | Index procedure until discharge
  Devices use

CONTACTS AND LOCATIONS:
Overall Officials: Deloose Koen, Dr, Study Chair — AZ Saint Blasius, Dendermonde, Belgium
Locations (17):
- LKH Univ.-Klinikum Graz, Ambulanz für Angiologie, Graz, Austria
- Belgium (5):
  - Ziekenhuis Oost Limburg, Genk, Genk
  - OLV Ziekenhuis Aalst, Aalst
  - A.Z. Sint-Blasius, Dendermonde
  - University Hospital Ghent, Ghent
  - vzw AZ Groeninge, Kortrijk
- Hopital Paris Saint Joseph, Paris, France
- Germany (3):
  - Universitätsklinikum Tübingen, Tübingen, Tübingen
  - Karolinen-Hospital, Klinikum Arnsberg, Arnsberg
  - Sank Gertrauden-Krankenhaus, Berlin
- Semmelweis University Hospital, Budapest, Hungary
- Italy (3):
  - Policlinico Abano Terme, Abano Terme, Abano Terme
  - Azienda Usl Toscana sud est, Arezzo, Arezzo
  - ospedaliero-universitaria Senese, Siena
- Hospital General de Guadalajara, Guadalajara, Spain
- Switzerland (2):
  - Ospedale Regionale di Lugano, Lugano, Lugano
  - KS Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD) is not yet drafted. No decision is taken to share it yet.